CLINICAL TRIAL: NCT02465034
Title: Noninvasive Brain Stimulation to Evaluate Neural Plasticity After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment and study activities were suspended due to COVID-19.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael R Borich, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00081268
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Cerebrovascular Stroke
Keywords: Neural plasticity; Noninvasive brain stimulation; Motor cortex
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Subcortical stroke (Active Comparator): Subjects with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function will undergo noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation will also be used which will be one of the following, a traditional or a corticocortical or a sham paired associative stimulation protocol. The subjects will also undergo median nerve stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation; Device: Traditional Paired Associative Stimulation; Device: Median Nerve Stimulation; Device: Corticocortical Paired Associative Stimulation; Device: Sham Paired Associative Stimulation
- Healthy Control (Active Comparator): Healthy individuals will undergo noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation will also be used which will be one of the following, a traditional or a corticocortical or a sham paired associative stimulation protocol.
  Interventions: Device: Transcranial Magnetic Stimulation; Device: Traditional Paired Associative Stimulation; Device: Median Nerve Stimulation; Device: Corticocortical Paired Associative Stimulation; Device: Sham Paired Associative Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) will be performed using the Magstim BiStim^2 paired pulse stimulator to measure transient cortical excitability. Single pulse transcranial magnetic stimulation applied at low frequencies (not greater than 0.25 hertz (Hz)) will be used. The may be repeated at multiple study visits. All five study visits will be completed within four weeks of the initial visit.
  Other Names: Magstim BiStim^2
Device: Traditional Paired Associative Stimulation — Paired associative stimulation (PAS) is a combination of transcranial magnetic stimulation (TMS) and electrical stimulation of the median nerve. 180 paired stimuli are delivered at 0.25 Hz for 12 minutes. Median nerve stimuli at 300% of the perceptual threshold will be applied 25ms prior to transcranial magnetic stimulation delivery over the ipsilesional (stroke) or non-dominant (control) cortex. Transcranial Magnetic Stimulation (TMS) will be performed using the Magstim BiStim^2 paired pulse stimulator unit and a bipolar bar electrode will be used for median nerve stimulation. This traditional paired associative stimulation may be repeated at multiple study visits. All five study visits will be completed within four weeks of the initial visit.
  Other Names: Magstim BiStim^2
Device: Median Nerve Stimulation — Stimulation of the median nerve will be performed using a bipolar bar electrode affixed to palmar aspect of the forearm proximal to the crease of the wrist bilaterally. Stimuli will be delivered 23ms prior to the transcranial magnetic stimulation (TMS) pulse with 0.1 milliseconds (ms) rectangular pulses at an intensity to evoke a 1 millivolt (mV) response in the abductor pollicis brevis (APB) muscle. This may may be repeated at multiple study visits. All five study visits will be completed within four weeks of the initial visit.
Device: Corticocortical Paired Associative Stimulation — Cortico-cortical Paired Associative Stimulation (CC-PAS) is a combination of TMS and electrical stimulation of the median nerve. 180 paired stimuli are delivered at 0.25 Hz for 12 minutes. The interstimulus interval will range from 5-15 ms depending on site of stimulation.TMS will be performed using the Magstim BiStim^2 paired pulse stimulator unit and a bipolar bar electrode will be used for median nerve stimulation. This CC-PAS may be repeated at multiple study visits. All five study visits will be completed within four weeks of the initial visit.
  Other Names: Magstim BiStim^2
Device: Sham Paired Associative Stimulation — The sham PAS is a combination of TMS and electrical stimulation of the median nerve. The coil is rotated and separated from the head with a plastic spacer to ensure indirect contact with the head.180 paired stimuli are delivered at 0.25 Hz for 12 minutes. TMS will be performed using the Magstim BiStim^2 paired pulse stimulator unit and a bipolar bar electrode will be used for median nerve stimulation. This sham paired associative stimulation may be repeated at multiple study visits. All five study visits will be completed within four weeks of the initial visit.
  Other Names: Magstim BiStim^2

SUMMARY:
The purpose of this study is to examine how different areas in the brain interact with each other and how using brain imaging and brain stimulation approaches can influence these interactions.

DETAILED DESCRIPTION:
Subcortical strokes affect small vessels deep in the brain, and typically present with motor hemiparesis. The investigator will assess the effects of Transcranial Magnetic Stimulation (TMS) on motor function and examine how different areas in the human brain interact with each other using brain imaging and brain stimulation. The investigator will also evaluate the capacity for noninvasive stimulation to transiently modify brain activity supporting arm movement.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-85 years
2. Middle cerebral artery stroke
3. Individuals with a first time stroke that affects the corona radiata and/or internal capsule

Exclusion Criteria:

1. Age outside the age range of 18-85 years
2. Signs of dementia (score < 24 on the Montreal Cognitive Assessment)
3. Aphasia (score < 13 on the Frenchay Aphasia Screen)
4. History of head trauma
5. History of a major psychiatric diagnosis
6. History of a neurodegenerative disorder
7. History of substance abuse
8. Contraindications to Transcranial Magnetic Stimulation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borich, DPT, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borich MR, Wolf SL, Tan AQ, Palmer JA. Targeted Neuromodulation of Abnormal Interhemispheric Connectivity to Promote Neural Plasticity and Recovery of Arm Function after Stroke: A Randomized Crossover Clinical Trial Study Protocol. Neural Plast. 2018 Mar 12;2018:9875326. doi: 10.1155/2018/9875326. eCollection 2018. PMID 29721010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began in May 2015 and all study follow up was completed by July 24, 2019. Study activities took place at the Emory Wesley Woods Health Center in Atlanta, Georgia.
Pre-assignment Details: Forty-five individuals gave consent to participate in the study and were enrolled into the appropriate study arm based on health status. Four screen failed or withdrew resulting in 41 who participated in the study. Participants with subcortical stroke could take part in both the PAS and CC-PAS studies.
Groups:
- Participants With Subcortical Stroke: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function undergoing noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation was used where participants received traditional PAS and sham PAS or a cortico-cortical paired associative stimulation (CC-PAS) and sham CC-PAS. Participants also underwent median nerve stimulation.
- Healthy Controls: Healthy individuals underwent noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation was used where participants received traditional PAS and sham PAS.
Period: Overall Study
Arm/Group | Participants With Subcortical Stroke | Healthy Controls
Started | 19 | 26
Started PAS | 12 | 21
Completed PAS | 9 | 20
Started CC-PAS | 16 | 0
Completed CC-PAS | 16 | 0
Completed | 16 | 20
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Screen fail | 2 | 0
Not completed — Could not be scheduled for study visit | 0 | 5

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes all individuals who consented to participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Subcortical Stroke | Healthy Controls | Total
Number analyzed (Participants) | 19 | 26 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (12.1) | 26.3 (6.1) | 39.9 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 25 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 26 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Long-term Potentiation-like Plasticity
Description: Long-term potentiation-like plasticity was measured using paired associative stimulation (PAS). PAS consists of repeated peripheral electric stimulation paired with Transcranial Magnetic Stimulation (TMS) applied to the motor cortex at varying interstimulus intervals. Participants received 180 paired stimuli at 0.25 hertz (Hz) for 12 minutes. Impaired long-term potentiation-like plasticity points towards reduced excitatory synaptic connectivity and deficits in sensorimotor integration. Decrease or no change in the amplitudes of motor-evoked potentials (MEPs) indicates impaired long-term potentiation-like plasticity.
Time Frame: Baseline, 1 Minute Post-Paired Associative Stimulation
Population: This analysis includes participants with complete and usable data. Errors with data acquisition occurred with three participants in the stroke PAS assessment, two participants in the stroke CC-PAS assessment, and three healthy controls. Two additional control participants were not included in the analysis due to data quality issues.
Measure: Mean (Standard Deviation); unit: microvolts (µV)
Groups:
- Subcortical Stroke PAS: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function receiving paired associative stimulation (PAS). PAS is a combination of transcranial magnetic stimulation (TMS) and electrical stimulation of the median nerve. 180 paired stimuli are delivered at 0.25 Hz for 12 minutes. Median nerve stimuli at 300% of the perceptual threshold is applied 25ms prior to transcranial magnetic stimulation delivery over the ipsilesional (stroke) or non-dominant (control) cortex.
- Subcortical Stroke PAS Sham: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function receiving sham paired associative stimulation (PAS).
- Subcortical Stroke CC-PAS: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function receiving cortico-cortical paired associative stimulation (CC-PAS). CC-PAS is a combination of TMS and electrical stimulation of the median nerve. 180 paired stimuli are delivered at 0.25 Hz for 12 minutes. The interstimulus interval ranges from 5-15 ms depending on site of stimulation.
- Subcortical Stroke CC-PAS Sham: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function receiving sham cortico-cortical paired associative stimulation (CC-PAS).
- Healthy Control Group: Healthy participants received noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation was also used.
- Healthy Control Sham: Healthy participants receiving sham paired associative stimulation (PAS).
Arm/Group | Subcortical Stroke PAS | Subcortical Stroke PAS Sham | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham | Healthy Control Group | Healthy Control Sham
Number analyzed (Participants) | 6 | 6 | 14 | 14 | 15 | 15
microvolts (µV)
  Baseline | 813.86 (619.81) | 819.47 (387.37) | 665.14 (645.05) | 427.80 (360.45) | 1408.08 (871.52) | 1025.60 (451.76)
  1 minute post-PAS | 1455.77 (1383.06) | 883.74 (424.24) | 644.46 (627.70) | 525.34 (502.67) | 1777.57 (1192.83) | 1121.38 (641.96)

2. Primary Outcome: Electroencephalography Recordings at Baseline and 5 MInutes Post-PAS
Description: Electroencephalography (EEG) data were recorded using a 64-channel TMS-compatible electrode cap (Easy Cap). Signals were collected at 2000 hertz (Hz) during pre- and post-transcranial magnetic stimulation epochs (-100ms to 200ms). Up to fifty suprathreshold (120% AMT) transcranial magnetic stimulation pulses were applied to motor cortex while the subject was seated quietly with eyes open. This procedure was conducted bilaterally. Data epochs (-1000 to 4000 ms with respect to TMS delivery) were extracted for subsequent imaginary phase coherence analysis. Post-TMS coherence values between electrodes overlying M1 bilaterally (C3 and C4) were calculated within the beta frequency range (15 to 30 Hz). EEG data values are unit-free that can range from 0 to 1. Higher values represent greater coherence which is thought to indicate stronger connectivity.
Time Frame: Baseline, 5 Minutes Post-Paired Associative Stimulation
Population: Only participants receiving CC-PAS were studied for this outcome. Errors with data acquisition occurred with two participants. Data were not collected for one participant due to EEG equipment malfunction, and not collected for one participant due to time constraints.
Measure: Mean (Standard Deviation); unit: coefficient of coherence
Arm/Group | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham
Number analyzed (Participants) | 12 | 12
coefficient of coherence
  Baseline | 0.20 (0.08) | 0.20 (0.07)
  5 minutes post-PAS | 0.19 (0.08) | 0.19 (0.07)

3. Primary Outcome: Abbreviated Wolf Motor Function Test Time
Description: Three items of the Wolf Motor Function Test (WMFT) were used to evaluate functional motor performance. The 3 items were selected based on task difficulty ranging from easiest (hand to table) to most difficult (stack checkers) along with a task of moderate difficulty (lift can). Each task has different control demands and number of actions required to complete successfully. Task performance is timed in seconds, with a maximum time of 120 seconds.
Time Frame: Baseline, 10 Minutes Post-Paired Associative Stimulation
Population: Only participants receiving CC-PAS were studied for this outcome. Errors with data acquisition occurred with two participants.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham
Number analyzed (Participants) | 14 | 14
seconds
  Hand to Table Baseline | 1.34 (1.00) | 1.20 (0.94)
  Hand to Table 10 Minutes Post-PAS | 1.22 (1.04) | 0.98 (0.76)
  Stack Checkers Baseline | 3.72 (3.91) | 3.26 (2.56)
  Stack Checkers 10 Minutes Post-PAS | 3.03 (2.29) | 3.20 (2.26)
  Lift Can Baseline | 7.76 (4.60) | 6.17 (2.52)
  Lift Can 10 Minutes Post-PAS | 7.40 (4.47) | 7.19 (2.93)

4. Secondary Outcome: Wolf Motor Function Test
Description: The arm function in subjects in the subcortical stroke group was evaluated by the Wolf Motor Function Test (WMFT). The test consists of timed and functional tasks and has 17 items. It is composed of 3 parts: Time, functional ability and strength and includes 15 function-based tasks and 2 strength based tasks. Items 1-6 involve timed functional tasks, items 7-14 are measures of strength, and the remaining 9 items consist of analyzing movement quality when completing various tasks. The examiner will test the less affected upper extremity followed by the most affected side. Scores are based on time taken to complete each task. The median time to complete all tasks will be be used to evaluate motor function. Larger values indicate greater upper extremity motor dysfunction.
Time Frame: Baseline
Population: This analysis includes participants with subcortical stroke, during the active PAS and CC-PAS assessments. Errors with data acquisition occurred with three participants in the stroke PAS assessment and two participants in the stroke CC-PAS assessment. This test was not performed for three participants receiving CC-PAS due to time constraints.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Subcortical Stroke PAS | Subcortical Stroke CC-PAS
Number analyzed (Participants) | 6 | 11
seconds | 5.79 (10.74) | 23.30 (47.81)

5. Secondary Outcome: Abbreviated Wolf Motor Function Test Time
Description: Three items of the WMFT were used to evaluate functional motor performance. The 3 items were selected based on task difficulty ranging from easiest (hand to table) to most difficult (stack checkers) along with a task of moderate difficulty (lift can). Each task has different control demands and number of actions required to complete successfully. Task performance will be timed, with a maximum time of 120 seconds.
Time Frame: 30 minutes post-Paired Associative Stimulation, 24 hours post-Paired Associative Stimulation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Subcortical Stroke CC-PAS Sham: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function receiving cortico-cortical paired associative stimulation (CC-PAS).
Arm/Group | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham
Number analyzed (Participants) | 14 | 14
seconds
  Hand to Table 30 minutes post-PAS | 1.09 (0.89) | 1.06 (0.80)
  Hand to Table 24 hours post-PAS | 1.18 (0.79) | 1.20 (1.10)
  Stack Checkers 30 minutes post-PAS | 3.15 (2.49) | 2.84 (1.41)
  Stack Checkers 24 hours post-PAS | 3.45 (4.78) | 2.81 (2.39)
  Lift Can 30 minutes post-PAS | 7.23 (3.83) | 7.79 (5.33)
  Lift Can 24 hours post-PAS | 7.23 (3.46) | 6.28 (2.90)

6. Secondary Outcome: Long-term Potentiation-like Plasticity
Description: Long-term potentiation-like plasticity was measured using paired associative stimulation (PAS). PAS consists of repeated peripheral electric stimulation paired with Transcranial Magnetic Stimulation (TMS) applied to the motor cortex at varying interstimulus intervals. Participants receive 180 paired stimuli at 0.25 Hz for 12 minutes. Impaired long-term potentiation-like plasticity points towards reduced excitatory synaptic connectivity and deficits in sensorimotor integration. Decrease or no change in the amplitudes of motor-evoked potentials (MEPs) indicates impaired long-term potentiation-like plasticity.
Time Frame: 30 minutes post-Paired Associative Stimulation, 24 hours post-Paired Associative Stimulation
Population: This analysis includes participants with complete and usable data. Errors with data acquisition occurred with three participants in the stroke PAS assessment, two participants in the stroke CC-PAS assessment, and three healthy controls. Two additional control participants were not included in the analysis due to data quality issues. Data from one participant with subcortical stroke receiving CC-PAS was not able to be analyzed due to excessive noise in the signal.
Measure: Mean (Standard Deviation); unit: microvolts (µV)
Arm/Group | Subcortical Stroke PAS | Subcortical Stroke PAS Sham | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham | Healthy Control Group | Healthy Control Sham
Number analyzed (Participants) | 6 | 6 | 13 | 14 | 15 | 15
microvolts (µV)
  30 minutes post-PAS | 1162.76 (585.18) | 847.61 (421.28) | 532.66 (510.49) | 503.87 (472.50) | 1757.44 (960.64) | 1310.29 (684.84)
  24 hours post-PAS | 1176.71 (737.16) | 749.86 (352.13) | 424.17 (410.79) | 445.29 (438.84) | 1542.62 (1219.24) | 1387.98 (758.53)

7. Secondary Outcome: Electroencephalography Recordings at 30 Minutes and 24 Hours Post-PAS
Description: as for outcome 2
Time Frame: 30 minutes post-Paired Associative Stimulation, 24 hours post-Paired Associative Stimulation
Population: Only participants receiving CC-PAS were studied for this outcome. Errors with data acquisition occurred with two participants. Data were not collected for one participant due to EEG equipment malfunction and not collected for another participant due to time constraints.
Measure: Mean (Standard Deviation); unit: coefficient of coherence
Arm/Group | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham
Number analyzed (Participants) | 12 | 12
coefficient of coherence
  30 minutes post-PAS | 0.18 (0.13) | 0.18 (0.07)
  24 hours post-PAS | 0.18 (0.07) | 0.17 (0.06)

8. Secondary Outcome: Serial Reaction Time Task (SRTT) Performance
Description: The SRTT involves pressing a key that corresponds to a target square positioned on a screen in front of the participant as quickly and accurately as possible. The response time for repeated and random sequences evaluate SRTT performance and skill is measured as the difference in response times between repeated and random sequences. Lower response times indicate better performance and a larger positive difference in response times represents greater sequence-specific skill. Negative values represent better performance on random sequences compared to repeated sequences.
Time Frame: Baseline, 10 minutes post-PAS, 30 minutes post-PAS, and 24 hours post-PAS
Population: Errors with data acquisition occurred with three participants in the stroke PAS assessment, two participants in the stroke CC-PAS assessment, and three healthy controls. Two additional control participants were not included due to data quality issues. One participant with subcortical stroke receiving PAS and two receiving CC-PAS were unable to perform the task due to severe upper extremity motor impairment.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Subcortical Stroke PAS | Subcortical Stroke PAS Sham | Subcortical Stroke CC-PAS | Subcortical Stroke CC-PAS Sham | Healthy Control Group | Healthy Control Sham
Number analyzed (Participants) | 5 | 5 | 12 | 12 | 15 | 15
milliseconds (ms)
  Baseline | 805.00 (188.63) | 1030.26 (398.40) | 19.21 (54.01) | 13.02 (67.51) | 45.13 (43.68) | 52.30 (48.71)
  10 minutes post-PAS | 806.00 (155.60) | 838.12 (172.58) | -1.69 (142.72) | 28.38 (114.26) | 52.73 (53.43) | 57.50 (59.76)
  30 minutes post-PAS | 812.80 (192.42) | 788.40 (197.86) | 9.35 (36.69) | 3.99 (70.74) | 66.16 (63.71) | 61.61 (57.97)
  24 hours post-PAS | 726.00 (112.81) | 790.25 (199.97) | -14.21 (114.31) | 8.94 (81.99) | 83.41 (82.96) | 77.05 (51.59)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time the intervention began through the final follow up assessment (up to 4 weeks).
Groups:
- Participants With Subcortical Stroke: Participants with subcortical stroke in the chronic phase of recovery with mild-moderate impairment of arm function undergoing noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation will also be used which will be one of the following, a traditional or a corticocortical or a sham paired associative stimulation protocol. The subjects also underwent median nerve stimulation.
- Healthy Controls: Healthy individuals underwent noninvasive targeting of cortical locations by stereotactic neuronavigation using Transcranial Magnetic Stimulation (TMS), median nerve stimulation and arm motor function assessments. A paired associative stimulation (PAS) protocol using noninvasive stimulation was also used, which was either a traditional or a corticocortical or a sham paired associative stimulation protocol.
Arm/Group | Participants With Subcortical Stroke | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/26
Other Adverse Events (participants affected / at risk) | 0/19 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT02465034/Prot_SAP_000.pdf